CLINICAL TRIAL: NCT03950050
Title: Ambroxol Therapy for Patients With Type 1 Gaucher Disease and Suboptimal Response to Enzyme Replacement Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0005-18-SZMC
Record Dates: First submitted 2018-08-06; First posted 2019-05-15 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-05

CONDITIONS: Gaucher Disease, Type 1
MeSH Terms: conditions — Gaucher Disease | interventions — Ambroxol

STUDY DESIGN:
Intervention Model Description: The aim of this single arm, phase II study is to evaluate the efficacy and safety of adding ambroxol to patients with type 1 GD and suboptimal response to ERT.
  HYPOTHESIS The addition of ambroxol will improve the disease related symptoms and disease impact of patients with GD with suboptimal response to ERT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambroxol (Experimental): Ambroxol therapy will be dosed up to 600 mg/day divided to twice a day starting 150 mg for the first month, 300 mg for the following month and 600 mg for the following month.
  The study was conducted in accordance with the provisions of the Declaration of Helsinki, Good Clinical Practice guidelines, and local laws and regulations.
  Interventions: Drug: Ambroxol

INTERVENTIONS:
Drug: Ambroxol — Ambroxol Hydrochloride therapy will be dosed up to 600 mg/day divided to twice a day starting 150 mg for the first month, 300 mg for the following month and 600 mg for the following month.
  The study was conducted in accordance with the provisions of the Declaration of Helsinki, Good Clinical Practice guidelines, and local laws and regulations.
  Other Names: Ambroxol Hydrochloride

SUMMARY:
Ambroxol hydrochloride, an over-the-counter antitussive available in many markets , was identified as an interesting pharmacological chaperone. In addition to a mucolytic action, ambroxol has antioxidant and anti-inflammatory properties. Importantly, ambroxol therapy was found safe when given to pregnant women for prevention of neonatal respiratory distress syndrome .

Thus, ambroxol, an oral available drug on the market, may be a safe option for GD patients with potential disease-specific efficacy and should be expanded into a clinical trial using higher doses and placebo-controlled design. The investigators propose to start with a phase II study for patients with type 1 GD and suboptimal response to ERT. In addition the investigators plan to open an international registry of patients with GD currently receiving ambroxol (off study).

DETAILED DESCRIPTION:
Introduction:

Description of the Problem:

Enzyme replacement therapy (ERT) makes a significant impact on the clinical manifestations and quality of life of patients with Gaucher disease (GD) . The goals of therapy focus mainly on platelets, hemoglobin, spleen, liver, bones and growth parameters for children.

ERT is mostly effective in patients with type 1 GD; still some patients don't achieve normalization or near normalization of the therapeutic targets . Glucosylsphingosine (LysoGb1) is the most specific and sensitive, and hence is probably the best currently available GD biomarker. A level of LysoGB1 < 140 ng/ml is considered a marker for controlled GD (personal communication).

Patients with GD may also experience chronic fatigue that causes functional disability and adversely affects quality of life . The fatigue severity scale (FSS) is a 9-item tool; each item is scored on a scale from 1 to 7, with a mean score of 4 or higher considered to represent significant fatigue . Patients with GD have improvements in fatigue within 6 months of starting ERT, and that it may be among the first symptoms to show significant improvement. Using the FSS, no association was identified between fatigue and time on ERT (P = 0.57). In a survey of patients with Type 1 GD and physicians, patients ascribed greater importance to fatigue than other disease parameters, while physicians placed more emphasis on objective measures of visceral and hematologic disease manifestations.

B. Pharmacological chaperones:

The underlying pathology in GD is not only due to the lysosomal accumulation of glucosylceramide in the tissue macrophages. There is a broader spectrum of lysosomal dysfunction and various intracellular and molecular changes that could lead to additional disease manifestations that are not affected by ERT. In particular, the retention of the mutant glucocerebrosidase within the endoplasmic reticulum (ER) which causes ER stress, unfolding protein response (UPR) and early ER associated degradation (ERAD) . These ER related changes are the rationale behind the use of pharmacological chaperones which are capable of partially removing the misfolded proteins from the ER, thereby relieving ER stress, avoiding ERAD and preventing consequent complications . Pharmacological chaperones increase glucocerebrosidase activity by stabilizing the enzyme in the lysosome.

C. The Therapy to be Examined:

Ambroxol hydrochloride, an over-the-counter antitussive available in many markets, was identified as an interesting pharmacological chaperone. In addition to a mucolytic action, ambroxol has antioxidant and anti-inflammatory properties . Importantly, ambroxol therapy was found safe when given to pregnant women for prevention of neonatal respiratory distress syndrome. In skin fibroblasts derived from Type 1 and Type 2 GD patients, ambroxol increases both the lysosomal fraction and the enzymatic activity of several mutant glucocerebrosidase variants with low toxicity . Incubation of human induced pluripotent stem cell macrophages from patients with type I-III GD with ambroxol corrected the abnormal phenotypes of GD macrophages. Ambroxol, has a small molecule chaperone, has been shown in healthy nonhuman primates to cross the blood-brain barrier, and increase brain glucocerebrosidase activity . In Drosophila neuropathic model, ambroxol was show to alleviate the neuronopathic phenotype through reducing ER stress ].

The investigators have performed a pilot study to test the tolerability and efficacy of ambroxol as a pharmacological chaperone in patients with symptomatic, type 1 GD who present with measurable disease parameters but are not receiving ERT in order to provide proof of concept and/or ascertain the suitability of ambroxol for a larger clinical trial [29] . The Israeli Ministry of Health Form 29c was employed to prescribe ambroxol for off-label use. Twelve patients were dispensed 2 capsules of 75 mg of ambroxol daily for 6 months. One patient withdrew because of a hypersensitivity reaction, one because of elective splenectomy. No patient experienced clinically relevant deterioration in disease parameters measured. One patient achieved a robust response relative to baseline: +16.2% hemoglobin; +32.9% platelets; -2.8% liver volume; and -14.4% spleen volume. Three patients elected to continue on ambroxol for a further 6 months: hemoglobin levels and liver volumes were relatively stable, but platelet counts further increased in the above patient (+52.6% from baseline) and spleen volumes decreased further in all three patients (-6.4%, -18.6%, and -23.4% from baseline) . More recently, a pilot study of ambroxol was done in five patients with neuronopathic GD in combination with enzyme replacement therapy [30]. High-dose oral Ambroxol had good safety and tolerability with clinical and laboratory signs of activity.

Thus, ambroxol, an oral available drug on the market, may be a safe option for GD patients with potential disease-specific efficacy and should be expanded into a clinical trial using higher doses and placebo-controlled design [31]. The investigators propose to start with a phase II study for patients with type 1 GD and suboptimal response to ERT. In addition the investigators plan to open an international registry of patients with GD currently receiving ambroxol (off study).

ELIGIBILITY:
Inclusion Criteria:

*Adult patients ≥ 18 years with type 1 GD and suboptimal response to ERT defined as one or more than one of the following: platelet count < 100 x 103/mm3 bone mineral density < -2 T score Lyso-GB1 > 200 ng/ml.

*No change in dose or preparation of ERT in the last 12 months (Except for Naive patients)

Exclusion Criteria:

* Patients with comorbidity that may impact on the primary and/or secondary endpoint.
* Pregnant women will be excluded from the study.
* Inability to cooperate with the study procedure
* Hypersensitivity or any other contraindication listed in the local labeling of ambroxol
* Refusal of patients to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Platelets count | 12 months.
  Increase in platelet count
bone mineral density evaluated by Dual Energy X-ray Absorptiometry (DEXA) | 12 months.
  Bone Mineral Densitometry (BMD)
Lyso-GB1 biomarker for Gaucher disease | 12 months
  decrease in Lyso-GB1.

SECONDARY OUTCOMES:
Patient-reported outcomes (PRO) | 12 months
  Improve in PRO from baseline
Fatigue Severity Scale (FSS) | 12 months
  Improve in FSS from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, Principal Investigator — Ari Zimran - Shaare Zedek
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ishay Y, Zimran A, Szer J, Dinur T, Ilan Y, Arkadir D. Combined beta-glucosylceramide and ambroxol hydrochloride in patients with Gaucher related Parkinson disease: From clinical observations to drug development. Blood Cells Mol Dis. 2018 Feb;68:117-120. doi: 10.1016/j.bcmd.2016.10.028. Epub 2016 Nov 12. PMID 27866808